CLINICAL TRIAL: NCT06858202
Title: Quality Improvement Project to Address Post Operative Distress and Pain for Patients Undergoing Surgery for Intra-Abdominal Malignancies
Brief Title: Study to Determine How Different Types of Coping Strategies Can Help People Manage Pain and Distress After Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Erin Ward, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 166993
Record Dates: First submitted 2025-02-21; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Psychological Distress; Intra-abdominal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Video-based Guided Mindfulness (Experimental): A 15-20-minute video based on previously tested and documented standards for guided meditation aimed at addressing pain and distress.
  Interventions: Behavioral: Mindfulness Intervention
- Video-based Guided Expressive Writing (Experimental): A 15-20-minute video based on expressive writing prompts aimed at addressing pain and distress. If the patient is assigned expressive writing, they will be offered a blank journal to use for the expressive writing interventions after randomization.
  Interventions: Behavioral: Mindfulness Intervention
- Non-Mindfulness Based Therapeutic Approaches (Active Comparator): Standard inpatient and outpatient resources available for Huntsman Cancer Institute patients through social work and the Wellness and Integrative Health Center. Participants will be encouraged to ask their providers for more information or if appropriate more consults to the appropriate resources if interested.
  Interventions: Behavioral: Non-mindfulness Intervention

INTERVENTIONS:
Behavioral: Mindfulness Intervention — Guided meditation or guided expressive writing
  Arms: Video-based Guided Expressive Writing; Video-based Guided Mindfulness
Behavioral: Non-mindfulness Intervention — Standard inpatient and outpatient resources available for Huntsman Cancer Institute patients through social work and the Wellness and Integrative Health Center. Participants will be encouraged to ask their providers for more information or if appropriate more consults to the appropriate resources if interested.
  Arms: Non-Mindfulness Based Therapeutic Approaches

SUMMARY:
The purpose of this study is to determine if different video based coping strategies can help patients undergoing surgery for cancer can improve patients pain and distress after surgery for their cancer.

The main questions this study aims to answer are:

* Is it possible to use video-based coping strategies to help manage pain and distress after surgery?
* Is one type of coping strategy better than another?

Researchers will compare mindfulness-based coping strategies (e.g., guided meditation, expressive writing, etc.) with non-mindfulness coping strategies (e.g., support from social workers and the wellness center, health education, etc.) to understand how these can help in post-surgery recovery, pain management, and distress.

Participants will:

* Provide their full name, date of surgery, e-mail address, and phone number and agree to be contacted via email or text messaging.
* Fill out some questionnaires before surgery, which should take 10-15 minutes.
* Be assigned to one of three coping strategies.
* Review a video (about 15-20 minutes long) or links to online resources before surgery and respond to questions about pain and distress before and after viewing these materials.
* Review additional videos or links 2, 3, and 4 days after surgery and respond to questions about pain and distress before and after viewing these materials.
* Complete additional questionnaires 2 weeks, 3 months, and 6 months after surgery. These questionnaires will be sent by text or email and should take about 10-15 minutes to complete.

DETAILED DESCRIPTION:
We propose to conduct a quality improvement project to determine the impact of different types of psychosocial support for patients undergoing surgery for intrabdominal malignancies.

This project will consist of a program evaluation/quality improvement study of existing pain and psychosocial management programs within the University of Utah Hospital System, which currently employs Study staff to provide mindfulness and non-mindfulness interventions for patients preparing for surgery and recovering from surgery. We wish to evaluate the differential impact of mindfulness interventions (e.g., guided meditation, expressive writing, etc.) and non-mindfulness interventions (. g., cognitive-behaviorally based psychoeducation, health education, grounding/earthing, and sham grounding/earthing, etc., support via social work and the wellness center, etc.) by randomly assigning patients to one of these approaches.

Objectives:

Aim 1 To assess the feasibility and acceptability of an application-based mindfulness or expressive writing intervention designed to address post-operative pain and distress, such as anxiety or depression, for patients undergoing surgery for intrabdominal malignancies.

Hypotheses: Greater than 50% of patients assigned to a mindfulness intervention, either guided meditation or expressive writing, will engage with at least one intervention, and over 30% of patients will engage with all four interventions.

Aim 2 To assess the differential effects of mindfulness vs. non-mindfulness therapeutic approaches on pain, distress, patient health engagement, and pain medication usage for patients preparing for/recovering from surgery for intraabdominal malignancies and identify the most sensitive instruments to detect this change in this population.

Hypotheses: Mindfulness-based therapeutic approaches, including guided meditation and expressive writing, will decrease pain, distress, and pain medicine usage and increase patient health engagement significantly more than standard non-mindfulness-based therapeutic approaches. We predict narcotic requirements during the post-operative period, and patient-reported pain scores will be the most sensitive.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking males or females 18 or older within the University of Utah Hospital system being treated for an intrabdominal malignancy.
* Patients undergoing surgical treatment of cancer within the abdominal cavity.

Exclusion Criteria:

* Altered mental status due to delirium or pharmacological sedation as determined by a clinical assessment conducted by a study staff.
* Non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of delivering video based mindfulness interventions | From enrollment to 6 months post-enrollment.
  The frequency that patients start and complete at least one mindfulness intervention will be evaluated and compared to the other two cohorts. The frequency of engaging with and completing the interventions will be reported descriptively. The Chi2 for Fisher's will be used for exact test.

SECONDARY OUTCOMES:
Participant-reported Global Impression of Change | From enrollment to 6 months post-enrollment.
  Patient global impression for change will be assessed using the PCIG (Rampakakis, Ste-Marie, et al. 2015, Perrot and Lantéri-Minet 2019) questionnaire. The questionnaire includes two items in which patients rate the change in their activity limitations, symptoms, and emotions on a descriptive scale from "No Change" = 1 to "A great deal better" = 7 and a visual scale from "Much better" = 0 to "Much worse" = 10.
Participant-reported pain intensity | From enrollment to 6 months post-enrollment.
  Change in pain symptoms will be assessed using the PROMIS Scale v2.0 Pain Intensity 3a questionnaire. This measure includes three items rating pain from "Had no pain" = 1 to "Very severe" = 5.
Participant-reported pain interference | From enrollment to 6 months post-enrollment.
  Change in pain interference will be assessed using the PROMIS Scale v1.1 Pain Interference 4a questionnaire. This measure includes three items rating the scale in which pain interferes with daily life from "Not at all" = 1 to "Very much" = 5.
Participant-reported physical function | From enrollment to 6 months post-enrollment.
  Change in physical will be assessed using the PROMIS Scale v2.0 Physical Function Short Form 6b questionnaire. This measure includes six items rating difficulty of daily tasks related to physical function from "Without any difficulty" = 1 to "Unable to do" = 5.
Participant-reported health engagement | From enrollment to 6 months post-enrollment.
  Participant health engagement will be assessed using the PHE questionnaire (Graffigna et. al 2015). This measure includes nine items in which patients rate how they feel about and engage with their disease. This scale has been adapted for study use to be rated on a scale from "never" = 1 to "always" = 5.
Participant-reported depression | From enrollment to 6 months post-enrollment.
  Change in emotional distress symptoms for depression will be assessed using the PROMIS Scale v1.0 Emotional Distress-Depression Short form 6a questionnaire. The questionnaire includes six items rating occurrence of different depression related emotions from "Never" = 1 to "Always" = 5.
Participant-reported anxiety | From enrollment to 6 months post-enrollment.
  Change in emotional distress symptoms for anxiety will be assessed using the PROMIS Scale v1.0 Emotional Distress-Anxiety Short form 6a questionnaire. The questionnaire includes six items rating occurrence of different anxiety related emotions from "Never" = 1 to "Always" = 5.
Participant-reported social isolation | From enrollment to 6 months post-enrollment.
  Change in levels of social isolation will be assessed using the PROMIS Scale v2.0 Social Isolation Short form 4a questionnaire. The questionnaire includes four items rating the occurrence of different feelings regarding social isolation from "Never" = 1 to "Always" = 5.
Participant-reported quality of life | From enrollment to 6 months post-enrollment.
  Participant quality of life will be assessed using the World Health Organization Quality of Life questionnaire. This questionnaire consists of two items that assess how patients feel about their quality of life on a scale from "Very poor" and "Very dissatisfied" =1 to "Very good" and "Very satisfied" = 5.
Participant use of pain medicine | From enrollment to 6 months post-enrollment.
  Patient narcotic consumption in the post-operative period will be collected via chart abstraction. Use of pain medicine will be compared with intervention acceptability and frequency of use at the end of the study, which may help guide future studies.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Health, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang R, Li L, Xu J, Ding ZT, Qiao J, Redding SR, Xianyu YY, Ouyang YQ. Effects of Structured Expressive Writing on Quality of Life and Perceived Self-Care Self-Efficacy of Breast Cancer Patients Undergoing Chemotherapy in Central China: A Randomized Controlled Trial. Healthcare (Basel). 2022 Sep 14;10(9):1762. doi: 10.3390/healthcare10091762. PMID 36141374
- [Background] Day MA, Ward LC, Ehde DM, Thorn BE, Burns J, Barnier A, Mattingley JB, Jensen MP. A Pilot Randomized Controlled Trial Comparing Mindfulness Meditation, Cognitive Therapy, and Mindfulness-Based Cognitive Therapy for Chronic Low Back Pain. Pain Med. 2019 Nov 1;20(11):2134-2148. doi: 10.1093/pm/pny273. PMID 30605517
- [Background] Rouleau CR, Garland SN, Carlson LE. The impact of mindfulness-based interventions on symptom burden, positive psychological outcomes, and biomarkers in cancer patients. Cancer Manag Res. 2015 Jun 1;7:121-31. doi: 10.2147/CMAR.S64165. eCollection 2015. PMID 26064068
- [Background] Hanley AW, Gililland J, Erickson J, Pelt C, Peters C, Rojas J, Garland EL. Brief preoperative mind-body therapies for total joint arthroplasty patients: a randomized controlled trial. Pain. 2021 Jun 1;162(6):1749-1757. doi: 10.1097/j.pain.0000000000002195. PMID 33449510
- [Background] Garland EL, Baker AK, Larsen P, Riquino MR, Priddy SE, Thomas E, Hanley AW, Galbraith P, Wanner N, Nakamura Y. Randomized Controlled Trial of Brief Mindfulness Training and Hypnotic Suggestion for Acute Pain Relief in the Hospital Setting. J Gen Intern Med. 2017 Oct;32(10):1106-1113. doi: 10.1007/s11606-017-4116-9. Epub 2017 Jul 12. PMID 28702870
- [Background] Zgierska AE, Burzinski CA, Cox J, Kloke J, Stegner A, Cook DB, Singles J, Mirgain S, Coe CL, Backonja M. Mindfulness Meditation and Cognitive Behavioral Therapy Intervention Reduces Pain Severity and Sensitivity in Opioid-Treated Chronic Low Back Pain: Pilot Findings from a Randomized Controlled Trial. Pain Med. 2016 Oct;17(10):1865-1881. doi: 10.1093/pm/pnw006. Epub 2016 Mar 10. PMID 26968850
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Rampakakis E, Ste-Marie PA, Sampalis JS, Karellis A, Shir Y, Fitzcharles MA. Real-life assessment of the validity of patient global impression of change in fibromyalgia. RMD Open. 2015 Sep 14;1(1):e000146. doi: 10.1136/rmdopen-2015-000146. eCollection 2015. PMID 26535150
- [Background] Perrot S, Lanteri-Minet M. Patients' Global Impression of Change in the management of peripheral neuropathic pain: Clinical relevance and correlations in daily practice. Eur J Pain. 2019 Jul;23(6):1117-1128. doi: 10.1002/ejp.1378. Epub 2019 Mar 18. PMID 30793414
- [Background] Hanley AW, Garland EL. Clarity of mind: Structural equation modeling of associations between dispositional mindfulness, self-concept clarity and psychological well-being. Pers Individ Dif. 2017 Feb 1;106:334-339. doi: 10.1016/j.paid.2016.10.028. Epub 2016 Nov 9. No abstract available. PMID 28584390
- [Background] Hanley AW, Garland EL. Dispositional Mindfulness Co-varies with Self-Reported Positive Reappraisal. Pers Individ Dif. 2014 Aug 1;66:146-152. doi: 10.1016/j.paid.2014.03.014. PMID 24904191
- [Background] Milbury K, Spelman A, Wood C, Matin SF, Tannir N, Jonasch E, Pisters L, Wei Q, Cohen L. Randomized controlled trial of expressive writing for patients with renal cell carcinoma. J Clin Oncol. 2014 Mar 1;32(7):663-70. doi: 10.1200/JCO.2013.50.3532. Epub 2014 Jan 27. PMID 24470003
- [Background] Carlson LE, Tamagawa R, Stephen J, Drysdale E, Zhong L, Speca M. Randomized-controlled trial of mindfulness-based cancer recovery versus supportive expressive group therapy among distressed breast cancer survivors (MINDSET): long-term follow-up results. Psychooncology. 2016 Jul;25(7):750-9. doi: 10.1002/pon.4150. Epub 2016 May 18. PMID 27193737
- [Background] Sanders SH, Harden RN, Vicente PJ. Evidence-based clinical practice guidelines for interdisciplinary rehabilitation of chronic nonmalignant pain syndrome patients. Pain Pract. 2005 Dec;5(4):303-15. doi: 10.1111/j.1533-2500.2005.00033.x. PMID 17177763
- [Background] Wipplinger F, Holthof N, Andereggen L, Urman RD, Luedi MM, Bello C. Meditation as an Adjunct to the Management of Acute Pain. Curr Pain Headache Rep. 2023 Aug;27(8):209-216. doi: 10.1007/s11916-023-01119-0. Epub 2023 Jun 7. PMID 37285010
- [Background] Ghoneim MM, O'Hara MW. Depression and postoperative complications: an overview. BMC Surg. 2016 Feb 2;16:5. doi: 10.1186/s12893-016-0120-y. PMID 26830195
- [Background] Mo M, Jia P, Zhu K, Huang W, Han L, Liu C, Huang X. Financial toxicity following surgical treatment for colorectal cancer: a cross-sectional study. Support Care Cancer. 2023 Jan 11;31(2):110. doi: 10.1007/s00520-022-07572-8. PMID 36629938
- [Background] Cimpean A, David D. The mechanisms of pain tolerance and pain-related anxiety in acute pain. Health Psychol Open. 2019 Nov 29;6(2):2055102919865161. doi: 10.1177/2055102919865161. eCollection 2019 Jul-Dec. PMID 31827877
- [Background] Baxter J, Welsh H, Grayer J. Mindfulness-based interventions for cancer-related pain and depression: a narrative review of current evidence and future potential. Curr Opin Support Palliat Care. 2019 Jun;13(2):81-87. doi: 10.1097/SPC.0000000000000428. PMID 30973395
- [Background] Apkarian AV, Bushnell MC, Treede RD, Zubieta JK. Human brain mechanisms of pain perception and regulation in health and disease. Eur J Pain. 2005 Aug;9(4):463-84. doi: 10.1016/j.ejpain.2004.11.001. Epub 2005 Jan 21. PMID 15979027
- [Background] Adamczyk AK, Ligeza TS, Wyczesany M. The dynamics of pain reappraisal: the joint contribution of cognitive change and mental load. Cogn Affect Behav Neurosci. 2020 Apr;20(2):276-293. doi: 10.3758/s13415-020-00768-7. PMID 31950439
- [Background] Low CA, Bovbjerg DH, Ahrendt S, Alhelo S, Choudry H, Holtzman M, Jones HL, Pingpank JF Jr, Ramalingam L, Zeh HJ 3rd, Zureikat AH, Bartlett DL. Depressive Symptoms in Patients Scheduled for Hyperthermic Intraperitoneal Chemotherapy With Cytoreductive Surgery: Prospective Associations With Morbidity and Mortality. J Clin Oncol. 2016 Apr 10;34(11):1217-22. doi: 10.1200/JCO.2015.62.9683. Epub 2016 Feb 22. PMID 26903574
- [Background] Rosenberger PH, Jokl P, Ickovics J. Psychosocial factors and surgical outcomes: an evidence-based literature review. J Am Acad Orthop Surg. 2006 Jul;14(7):397-405. doi: 10.5435/00124635-200607000-00002. PMID 16822887
- [Background] Sharp L, Carsin AE, Timmons A. Associations between cancer-related financial stress and strain and psychological well-being among individuals living with cancer. Psychooncology. 2013 Apr;22(4):745-55. doi: 10.1002/pon.3055. Epub 2012 Mar 12. PMID 22411485
- [Background] Zhu J, Fang F, Sjolander A, Fall K, Adami HO, Valdimarsdottir U. First-onset mental disorders after cancer diagnosis and cancer-specific mortality: a nationwide cohort study. Ann Oncol. 2017 Aug 1;28(8):1964-1969. doi: 10.1093/annonc/mdx265. PMID 28525559
- [Background] Klaassen Z, Wallis CJD, Goldberg H, Chandrasekar T, Sayyid RK, Williams SB, Moses KA, Terris MK, Nam RK, Urbach D, Austin PC, Kurdyak P, Kulkarni GS. The impact of psychiatric utilisation prior to cancer diagnosis on survival of solid organ malignancies. Br J Cancer. 2019 Apr;120(8):840-847. doi: 10.1038/s41416-019-0390-0. Epub 2019 Mar 6. PMID 30837680
- [Background] Lee DS, Marsh L, Garcia-Altieri MA, Chiu LW, Awad SS. Active Mental Illnesses Adversely Affect Surgical Outcomes. Am Surg. 2016 Dec 1;82(12):1238-1243. PMID 28234191
- [Background] Graffigna G, Barello S, Bonanomi A, Lozza E. Measuring patient engagement: development and psychometric properties of the Patient Health Engagement (PHE) Scale. Front Psychol. 2015 Mar 27;6:274. doi: 10.3389/fpsyg.2015.00274. eCollection 2015. PMID 25870566